CLINICAL TRIAL: NCT06485479
Title: Identifying Effective Ads to Encourage Quitting Smoking Among People Who Smoke Menthol Cigarettes
Brief Title: Effective Ads for Quitting Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-2450; U54DA060049 (NIH)
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Smoking Behaviors
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Ads about response efficacy for quitting smoking (Experimental): Participants will view ads designed to increase response efficacy for quitting cigarettes.
  Interventions: Behavioral: Intervention ads
- Ads about self-efficacy for quitting smoking (Experimental): Participants will view ads designed to increase self-efficacy to quit smoking.
  Interventions: Behavioral: Intervention ads
- Ads about motivation to quit smoking (Experimental): Participants will view ads designed to increase motivation to quit smoking.
  Interventions: Behavioral: Intervention ads
- Ads about reading (Other): Participants will view non-smoking related ads on the benefits of reading.
  Interventions: Behavioral: Control ads
- Ads about passwords (Other): Participants will view non-smoking related ads on passwords.
  Interventions: Behavioral: Control ads

INTERVENTIONS:
Behavioral: Intervention ads — The ads will be on topics to encourage quitting smoking, formatted as multi-color text with graphic elements. Trial investigators developed the ads and optimized them to be readable when delivered in an SMS text message.
  Arms: Ads about motivation to quit smoking; Ads about response efficacy for quitting smoking; Ads about self-efficacy for quitting smoking
Behavioral: Control ads — The ads will be on topics unrelated to quitting smoking, formatted as black text on a white field. Trial investigators developed the ads and optimized them to be readable when delivered in an SMS text message.
  Arms: Ads about passwords; Ads about reading

SUMMARY:
The main purpose of this trial is to identify effective quit smoking ads for people who smoke menthol cigarettes. Investigators will conduct an online randomized trial with a nationally representative sample of ~1,400 US adults (ages 21+) who smoke menthol cigarettes.

DETAILED DESCRIPTION:
This trial will evaluate the effectiveness of efficacy-based quit smoking ads in a 5 (theme) x 6 (ad) mixed factorial randomized design.

Recruitment: A survey company will recruit ~1,400 participants. Participants will complete a screener to confirm that they are US adults (ages 21+), currently smoke menthol cigarettes, and are able to read and speak English. A portion of the sample will be nationally representative, and a portion will be a convenience sample.

Informed Consent: The consent form will appear on the first page of the survey. Participants will provide their consent to be in the trial by clicking on a button that forwards to the next page of the survey.

Randomization: After consent, the survey software will randomize participants to 1 of 5 themes between-subjects. The design will include 3 intervention ad themes about quitting smoking (self-efficacy ads, response efficacy ads, or motivation ads) and 2 control ad themes about neutral non-smoking related topics (reading or password safety).

Each participant will view 6 ads on their assigned theme, presented in a random order.

Assessment: Participants will complete a ~15 minute online survey one time.

ELIGIBILITY:
This national trial is not open to enrollment from the general public. Participation is restricted to individuals who meet the following inclusion and exclusion criteria:

Inclusion Criteria

* Currently smoke menthol cigarettes
* Be a member of the AmeriSpeak online survey panel or their convenience sample
* Live in the US
* Be age 21 years or older
* Read and speak English

Exclusion Criteria

* Not currently smoke menthol cigarettes
* Not be a member of the AmeriSpeak online survey panel or their convenience sample
* Not live in the US
* Be younger than age 21 years
* Not be able to read and speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1236 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noel Brewer, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Marissa G Hall, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The trial investigators will produce a de-identified dataset and codebook for sharing with external investigators, making use of the UNC Dataverse digital data repository (dataverse.unc.edu) hosted by the Odum Institute Data Archive.
Supporting Information: SAP
Time Frame: The data will be available beginning 12 and continuing for 36 months following the primary publication.
Access Criteria: To obtain a copy of the dataset and codebook, a research scientist will submit a request in writing, identifying themselves and their affiliated institution, indicating what they plan to do with the data, and including assurances that they will not share the data with others without the written permission of the PI. Requestors must already have institutional review board, independent ethics committee, or research ethics board approval, as applicable. Requestors must obtain a data use agreement through UNC's Office of Industry Contracting (OIC@unc.edu) to receive the dataset and codebook and agree to acknowledge NIH and the study investigators in any publications resulting from the data.

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ads About Response Efficacy for Quitting Smoking | Ads About Self-efficacy for Quitting Smoking | Ads About Motivation to Quit Smoking | Ads About Reading | Ads About Passwords
Started | 247 | 242 | 251 | 249 | 247
Completed | 247 | 242 | 251 | 249 | 247
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ads About Response Efficacy for Quitting Smoking | Ads About Self-efficacy for Quitting Smoking | Ads About Motivation to Quit Smoking | Ads About Reading | Ads About Passwords | Total
Number analyzed (Participants) | 247 | 242 | 251 | 249 | 247 | 1236
Age, Customized [Count of Participants; unit: Participants]
  21-29 years | 30 | 22 | 23 | 30 | 28 | 133
  30-39 years | 73 | 71 | 73 | 66 | 73 | 356
  40-49 years | 48 | 53 | 55 | 65 | 54 | 275
  50-59 years | 38 | 38 | 40 | 40 | 39 | 195
  60+ years | 58 | 58 | 60 | 48 | 53 | 277
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 162 | 156 | 160 | 150 | 777
  Male | 98 | 80 | 95 | 89 | 97 | 459
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 133 | 124 | 128 | 136 | 121 | 642
  Non-Hispanic Black | 59 | 66 | 69 | 54 | 63 | 311
  Hispanic | 26 | 27 | 35 | 41 | 37 | 166
  Multiracial | 15 | 8 | 7 | 7 | 10 | 47
  Another race / ethnicity | 14 | 17 | 12 | 11 | 16 | 70

OUTCOME MEASURES:

1. Primary Outcome: Perceived Message Effectiveness for Motivation
Description: Perceived effectiveness of the ads at encouraging quitting smoking, measured by 1 survey item for each ad (6 items total). Range 1 to 5, with higher values indicating higher perceived message effectiveness.
Time Frame: During exposure to the ads, assessed during one-time online 15-minute survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ads About Response Efficacy for Quitting Smoking | Ads About Self-efficacy for Quitting Smoking | Ads About Motivation to Quit Smoking | Ads About Reading | Ads About Passwords
Number analyzed (Participants) | 247 | 242 | 251 | 249 | 247
score on a scale | 3.18 (1.05) | 2.40 (0.99) | 2.49 (1.02) | 1.49 (0.87) | 1.41 (0.88)
Statistical Analysis 1: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Self-efficacy for Quitting Smoking; Test type: Superiority; p < .001, Regression, Linear
Statistical Analysis 2: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Motivation to Quit Smoking; Test type: Superiority; p < .001, Regression, Linear
Statistical Analysis 3: Comparison: Ads About Reading vs Ads About Passwords; Test type: Superiority; p = .56, Regression, Linear

2. Secondary Outcome: Perceived Message Effectiveness for Response Efficacy
Description: Perceived effectiveness of the ads at communicating the benefits of quitting smoking, measured by 1 survey item for each ad (6 items total). Range 1 to 5, with higher values indicating higher perceived message effectiveness.
Time Frame: During exposure to the ads, assessed during one-time online 15-minute survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ads About Response Efficacy for Quitting Smoking | Ads About Self-efficacy for Quitting Smoking | Ads About Motivation to Quit Smoking | Ads About Reading | Ads About Passwords
Number analyzed (Participants) | 247 | 242 | 251 | 249 | 247
score on a scale | 3.32 (1.01) | 2.23 (1.02) | 2.33 (1.04) | 1.48 (0.86) | 1.44 (0.91)
Statistical Analysis 1: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Self-efficacy for Quitting Smoking; Test type: Superiority; p < .001, Regression, Linear
Statistical Analysis 2: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Motivation to Quit Smoking; Test type: Superiority; p < .001, Regression, Linear
Statistical Analysis 3: Comparison: Ads About Reading vs Ads About Passwords; Test type: Superiority; p = .35, Regression, Linear

3. Secondary Outcome: Perceived Message Effectiveness for Self-efficacy
Description: Perceived effectiveness of the ads at creating confidence that one can quit smoking, measured by 1 survey item for each ad (6 items total). Range 1 to 5, with higher values indicating higher perceived message effectiveness.
Time Frame: During exposure to the ads, assessed during one-time online 15-minute survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ads About Response Efficacy for Quitting Smoking | Ads About Self-efficacy for Quitting Smoking | Ads About Motivation to Quit Smoking | Ads About Reading | Ads About Passwords
Number analyzed (Participants) | 247 | 242 | 251 | 249 | 247
score on a scale | 2.94 (1.14) | 2.49 (0.96) | 2.45 (1.04) | 1.48 (0.85) | 1.43 (0.89)
Statistical Analysis 1: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Self-efficacy for Quitting Smoking; Test type: Superiority; p < .001, Regression, Linear
Statistical Analysis 2: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Motivation to Quit Smoking; Test type: Superiority; p < .001, Regression, Linear
Statistical Analysis 3: Comparison: Ads About Reading vs Ads About Passwords; Test type: Superiority; p = .62, Regression, Linear

4. Secondary Outcome: Intentions to Quit Smoking
Description: Motivation to quit smoking, measured by 1 survey item. Range 1 to 5, with higher values indicating higher intentions to quit smoking.
Time Frame: After exposure to the ads, assessed during one-time online 15-minute survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ads About Response Efficacy for Quitting Smoking | Ads About Self-efficacy for Quitting Smoking | Ads About Motivation to Quit Smoking | Ads About Reading | Ads About Passwords
Number analyzed (Participants) | 247 | 242 | 251 | 249 | 247
score on a scale | 3.14 (1.21) | 2.90 (1.31) | 2.99 (1.29) | 2.94 (1.34) | 2.82 (1.35)
Statistical Analysis 1: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Self-efficacy for Quitting Smoking; Test type: Superiority; p = .03, Regression, Linear
Statistical Analysis 2: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Motivation to Quit Smoking; Test type: Superiority; p = .17, Regression, Linear
Statistical Analysis 3: Comparison: Ads About Reading vs Ads About Passwords; Test type: Superiority; p = .33, Regression, Linear

5. Secondary Outcome: Response Efficacy
Description: Belief that quitting smoking improves health, measured by 1 survey item. Range 1 to 5, with higher values indicating higher response efficacy.
Time Frame: After exposure to the ads, assessed during one-time online 15-minute survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ads About Response Efficacy for Quitting Smoking | Ads About Self-efficacy for Quitting Smoking | Ads About Motivation to Quit Smoking | Ads About Reading | Ads About Passwords
Number analyzed (Participants) | 247 | 242 | 251 | 249 | 247
score on a scale | 3.50 (0.79) | 3.93 (1.18) | 3.96 (1.12) | 4.00 (1.23) | 3.91 (1.25)
Statistical Analysis 1: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Self-efficacy for Quitting Smoking; Test type: Superiority; p < .001, Regression, Linear
Statistical Analysis 2: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Motivation to Quit Smoking; Test type: Superiority; p < .001, Regression, Linear
Statistical Analysis 3: Comparison: Ads About Reading vs Ads About Passwords; Test type: Superiority; p = .38, Regression, Linear

6. Secondary Outcome: Self-efficacy
Description: Confidence that one can quit smoking, measured by 1 survey item. Range 1 to 5, with higher values indicating higher self-efficacy.
Time Frame: After exposure to the ads, assessed during one-time online 15-minute survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ads About Response Efficacy for Quitting Smoking | Ads About Self-efficacy for Quitting Smoking | Ads About Motivation to Quit Smoking | Ads About Reading | Ads About Passwords
Number analyzed (Participants) | 247 | 242 | 251 | 249 | 247
score on a scale | 2.93 (1.27) | 2.87 (1.27) | 2.88 (1.19) | 2.87 (1.27) | 2.78 (1.29)
Statistical Analysis 1: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Self-efficacy for Quitting Smoking; Test type: Superiority; p = .6, Regression, Linear
Statistical Analysis 2: Comparison: Ads About Response Efficacy for Quitting Smoking vs Ads About Motivation to Quit Smoking; Test type: Superiority; p = .65, Regression, Linear
Statistical Analysis 3: Comparison: Ads About Reading vs Ads About Passwords; Test type: Superiority; p = .4, Regression, Linear

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent, through completion of ~15 minute one time online survey.
Arm/Group | Ads About Response Efficacy for Quitting Smoking | Ads About Self-efficacy for Quitting Smoking | Ads About Motivation to Quit Smoking | Ads About Reading | Ads About Passwords
All-Cause Mortality (participants affected / at risk) | 0/247 | 0/242 | 0/251 | 0/249 | 0/247
Serious Adverse Events (participants affected / at risk) | 0/247 | 0/242 | 0/251 | 0/249 | 0/247
Other Adverse Events (participants affected / at risk) | 0/247 | 0/242 | 0/251 | 0/249 | 0/247

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT06485479/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT06485479/ICF_001.pdf